CLINICAL TRIAL: NCT00393887
Title: Inguinal Hernia Study: A Double Blinded Randomized Prospective Study
Brief Title: Inguinal Hernia Study Using Biodesign IHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Collaborators: Cook Biotech Incorporated (Industry); MED Institute, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-28044; 05-003
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; polypropylene; Biodesign IHM; lichtenstein
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Biodesign IHM Graft placement
  Interventions: Device: Biodesign IHM
- 2 (Active Comparator): Polypropylene mesh placement
  Interventions: Device: Polypropylene mesh

INTERVENTIONS:
Device: Biodesign IHM — Biodesign IHM is placed to reinforce the hernia repair
  Other Names: SurgiSIS IHM
  Arms: 1
Device: Polypropylene mesh — Polypropylene mesh is used to reinforce the hernia repair.
  Arms: 2

SUMMARY:
Aim is to evaluate outcomes of inguinal hernia repair incorporating the standard Lichtenstein (open) repair using Biodesign IHM in a double blind (physician evaluator and patient will be blinded), randomized, prospective comparative study with polypropylene mesh. Primary outcome is recurrence at 1 year. Hernia recurrence will be confirmed via ultrasound or CT scan.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Diagnosis of Unilateral inguinal hernia repair
* Able to provide written consent

Exclusion Criteria:

* Incarcerated hernia
* Allergic or religious beliefs that disallow porcine material
* Previous hernia repair on the designated hernia site
* Class IV or V anesthesia requirements
* Bowel obstruction
* Peritonitis
* Life expectancy < 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Timmons, M.D., Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- See also: Biologic vs Synthetic Inguinal Hernia Repair: 1-year Results of a Randomized Double-Blinded Trial — http://www.ncbi.nlm.nih.gov/pubmed/24655865

RESULTS

PARTICIPANT FLOW:
Groups:
- Biodesign IHM Graft: Biodesign Inguinal Hernia Matrix (IHM)
- Polypropylene Mesh: Synthetic polypropylene mesh
Period: Overall Study
Arm/Group | Biodesign IHM Graft | Polypropylene Mesh
Started | 50 | 50
1 Year | 45 | 50
Completed | 34 | 41
Not Completed | 16 | 9
Not completed — Physician Decision | 5 | 0
Not completed — Lost to Follow-up | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biodesign IHM Graft | Polypropylene Mesh | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Full Range); unit: years] | 64 [24 to 85] | 59 [25 to 87] | 61.5 [24 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Inguinal Hernia Recurrence
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Biodesign IHM Graft: Inguinal hernia repair with Biodesign Inguinal Hernia Matrix (IHM)
- Polypropylene Mesh: Inguinal hernia repair with Polypropylene mesh
Arm/Group | Biodesign IHM Graft | Polypropylene Mesh
Number analyzed (Participants) | 45 | 50
participants | 3 | 0
Statistical Analysis 1: Comparison: Biodesign IHM Graft vs Polypropylene Mesh; Two-sided Fisher's exact test; Test type: Superiority or Other; p = 0.11, Fisher Exact

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Biodesign IHM Graft | Polypropylene Mesh
Serious Adverse Events (participants affected / at risk) | 7/45 | 5/50
Other Adverse Events (participants affected / at risk) | 18/45 | 15/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biodesign IHM Graft (N=45) | Polypropylene Mesh (N=50)
Hematoma requiring hospitalization (Vascular disorders) | 1 (1) | 0 (0) — unrelated to the device
Urinary tract infection (UTI) requiring hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0) — unrelated to the device
MI resulting in death (Cardiac disorders) | 1 (1) | 0 (0) — unrelated to the device
Scrotal hematoma requiring hospitalization (Vascular disorders) | 1 (1) | 0 (0) — unrelated to the device
Bradycardia during hernia repair (Cardiac disorders) | 1 (1) | 0 (0) — unrelated to the device
Right inguinal pain, inflammation, and tenderness (Infections and infestations) | 1 (1) | 0 (0) — Requiring hospitalization - possibly related to the device
Left groin pain and scrotal swelling (Infections and infestations) | 1 (1) | 0 (0) — Requiring hospitalization - possibly related to the device
Diverticulitis and prostatitis requiring hospitalization (Infections and infestations) | 0 (0) | 1 (1) — unrelated to the device
Substantial bleeding with central-line placement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — unrelated to the device
Motorcycle accident resulting in death (General disorders) | 0 (0) | 1 (1) — unrelated to the device
Severe pain requiring hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1) — unrelated to the device
Urinary retention requiring overnight observation (Renal and urinary disorders) | 0 (0) | 1 (1) — unrelated to the device
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biodesign IHM Graft (N=45) | Polypropylene Mesh (N=50)
Postoperative pain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Hematoma (Surgical and medical procedures) | 6 (6) | 1 (1)
Seroma (Surgical and medical procedures) | 5 (5) | 0 (0)
Neuralgia (Nervous system disorders) | 4 (4) | 6 (6)
Testicular problems (Renal and urinary disorders) | 5 (5) | 4 (4)
Urinary retention (Renal and urinary disorders) | 6 (6) | 3 (3)
Incisional pain (Surgical and medical procedures) | 2 (2) | 4 (4)
Surgical site reaction (Surgical and medical procedures) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days